CLINICAL TRIAL: NCT03487549
Title: A Phase 2, Open Label Study to Evaluate the Efficacy, Safety and Tolerability of VP-102 in Subjects With Common Warts (Verruca Vulgaris)
Brief Title: Cantharidin and Occlusion in Verruca Epithelium
Acronym: COVE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verrica Pharmaceuticals Inc. (Industry)
Collaborators: Instat Consulting, Inc. (Other); Paidion Research, Inc. (Industry); BioClinica, Inc. (Industry); ALMAC Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VP-102-105
Record Dates: First submitted 2018-03-21; First posted 2018-04-04 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2021-08

CONDITIONS: Common Wart; Warts Hand; Warts; Papillomavirus Infections; DNA Virus Infections; Skin Diseases, Viral; Skin Diseases, Infectious; Skin Diseases; Virus Diseases; Tumor Virus Infections; Verruca Vulgaris; Verruca
MeSH Terms: conditions — Warts; Papillomavirus Infections; DNA Virus Infections; Skin Diseases, Viral; Skin Diseases, Infectious; Skin Diseases; Virus Diseases; Tumor Virus Infections

STUDY DESIGN:
Intervention Model Description: This study has 2 cohorts. Cohort 1 of the study enrolled 21 subjects and has completed all subject related study activities. Analysis is to be conducted at Day 84. Cohort 2 will utilize 4 sites with an enrollment of approximately 35 subjects. The primary analysis will be conducted at Day 84 with an additional period of follow up out to Day 147.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- VP-102 (Experimental): Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator.
  Interventions: Combination Product: VP-102 Cantharidin topical film forming solution; Combination Product: VP-102 Cantharidin, topical film forming solution

INTERVENTIONS:
Combination Product: VP-102 Cantharidin topical film forming solution — VP-102, a single-use drug device combination product containing (cantharidin) topical solution, 0.7% (w/v). Treatment interval of at least 14 days between treatments.
  Other Names: VP-102-Cantharidin, film forming solution, VP-102 - Cohort 1
Combination Product: VP-102 Cantharidin, topical film forming solution — VP-102, a single-use drug device combination product containing (cantharidin) topical solution, 0.7% (w/v). Treatment interval of at least 21 days between treatments.
  Other Names: VP-102 Cantharidin, film forming solution, VP-102 - Cohort 2

SUMMARY:
This is a Phase 2, open label study (Study number VP-102-105; referred to as COVE-1 [Cantharidin and Occlusion in Verruca Epithelium]) to evaluate the efficacy, safety and tolerability of VP-102 treatment in subjects with common warts. This study has two Cohorts.

DETAILED DESCRIPTION:
The first Cohort (Cohort 1) utilizes a treatment interval of at least 14 days between treatments with longer treatment intervals being allowed depending on a specific patient's clinical response.Twenty Subjects (2 years and older) are targeted completing End of Study (EOS) visit in Cohort 1.

The second Cohort (Cohort 2) utilizes a treatment interval of 21 days between treatments. Paring of lesions is allowed. Approximately 35 subjects (12 years and older) will be enrolled in Cohort 2. Up to 4 sites will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be healthy, immunocompetent males or females at least 2 years of age and older for Cohort 1 and 12 years of age and older for Cohort 2.
2. Present with 1-6 common warts (verruca vulgaris) located anywhere on the body except for the following prohibited areas: the eye area (including eyelids), lips, oral cavity, nasal cavity, inside of the ears, palms of the hands, volar surface of the fingers or toes, under the finger nails (near and on the sides of the nails is allowed for Cohort 1, but warts near and on the sides of the nail (e.g., periungual) are not allowed in Cohort 2), soles of the feet, or the anogenital area. (Warts within 10 mm of a mucosal surface should not be treated).
3. Have warts that are ≤10 mm in diameter and ≤3 mm in height. (Subjects with warts that are adjacent, touching or clustered may be included so long as the combined diameter in the longest direction does not exceed 10 mm. Individual lesions that are adjacent, touching or clustered should be counted as distinct lesions for the purposes of tracking, inclusion and clearance)(subjects in Cohort 2 can be pared, when necessary and appropriate, prior to evaluating height eligibility) .
4. Have warts that have been present for at least 4 weeks at the time of the baseline visit.
5. Consent to having all warts treated (the physician must also be willing to treat all warts initially present).
6. Be otherwise medically healthy with no clinically significant medical history, physical examination or vital signs as determined by the investigator.
7. Be free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of Aes.
8. Refrain from swimming, bathing or prolonged immersion in water or any liquids until the Study drug is removed.
9. Have the ability, or have a guardian with the ability, to follow study instructions and be likely to complete all study requirements.
10. Agree to use no wart-removing product (prescription or over-the-counter [OTC]) other than the Study drug during the course of the study.
11. Provide written informed consent or assent in a manner approved by the institutional review board (IRB) and/or have a parent/guardian provide written informed consent as evidenced by the signature on an IRB approved assent/consent form.
12. Provide written authorization for use and disclosure of protected health information.
13. If participating in the optional photographic portion of the study, agree to allow photographs of warts to be taken at each Treatment Visit by the research team and agree to share photos taken at home with the research team via text, email or in-person upload.

Exclusion Criteria:

1. Are unable to cooperate with the requirements or visits of the study, as determined by the investigator.
2. Are systemically immunosuppressed or have required, or will require, systemic immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) within 30 days prior to enrollment or during the course of the study. (Routine use of inhaled or intranasal corticosteroids during the study is allowed)
3. Have any chronic or acute medical condition that, in the opinion of the investigator, may interfere with the study results or place the subject at undue risk. (e.g., human immunodeficiency virus, systemic lupus erythematosus, viral hepatitis, uncontrolled diabetes). NOTE: Immunizations and flu shots may be administered throughout the study, but not within 5 days before or after treatment.
4. Have more than 6 common warts at baseline.
5. Present with any verruca plana, mosaiform, filiform, subungual (under the nail), genital or anal warts. In Cohort 2, subjects with periungual warts are also excluded.
6. Have any warts present at baseline in an anatomic location that the subject, parent/guardian or the physician is unwilling to treat or are located in an area that cannot be easily occluded with tape.
7. Have had any previous treatment of common warts including, but not limited to, the use of cantharidin, antivirals, retinoids, salicylic acid, lactic acid, hydrogen peroxide, candida antigen, diphencyprone, dinitrochlorobenzene, sandalwood oil, thuja oil, squaric acid dibutyl ester, povidone iodine, nitric oxide, curettage or freezing of warts in the past 14 days. In addition, these treatments or any other over-the-counter wart treatment should not be implemented during the course of the study.
8. Have been treated within 14 days with a product that contains cantharidin (topical or homeopathic preparations) for any reason prior to screening.
9. Have received another investigational product as part of a clinical trial within 30 days prior to the first application of the Study drug.
10. Currently have or have a history of epidermodysplasia verruciformis.
11. Have a history of illness or any dermatologic disorder, which, in the opinion of the investigator, will interfere with accurate assessment of the warts or increase the risk of adverse events.
12. Have an active malignancy or are undergoing treatment for any malignancy.
13. Have a history or presence of clinically significant medical, psychiatric, or emotional condition or abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of the data.
14. Have a history or presence of hypersensitivity or an idiosyncratic reaction to the Study drug or related compounds, or drug product excipients (acetone, ethyl alcohol, nitrocellulose, hydroxypropyl cellulose, castor oil, camphor, gentian violet, and denatonium benzoate).
15. Have a condition or situation that may interfere significantly with the subject's participation in the study (e.g., subjects who required hospitalization in the 2 months prior to screening for an acute or chronic condition including alcohol or drug abuse), at the discretion of the investigator.
16. Are sexually active or may become sexually active and are unwilling to practice responsible birth control methods. (e.g., combination of condoms and foam, birth control pills, intrauterine device, patch, shot and vaginal ring, etc.). Withdrawal is not an acceptable method of birth control. Females that have reached menarche must have a negative urine pregnancy test at each visit prior to treatment with Study drug.
17. Are pregnant or breastfeeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Nasir, MD, Principal Investigator — Cohort 1: Wake Dermatology; Scott Guenthner, MD, Principal Investigator — Cohort 2: Indiana Clinical Trials Center
Locations (5):
- United States (5):
  - Cohort 2: Applied Research Center of Arkansas, Little Rock, Arkansas
  - Cohort 2: Solutions Through Advanced Research, Jacksonville, Florida
  - Cohort 2: The Indiana Clinical Trials Center, Plainfield, Indiana
  - Cohort 2: Clarkston Skin Research, Clarkston, Michigan
  - Cohort 1-Wake Research Associates, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guenthner S, McFalda W, Kwong P, Eads K, McCafferty M, Rieger J, Glover DK, Willson C, Burnett P, Olivadoti M. COVE-1: A Phase 2, Open-Label Study to Evaluate Efficacy and Safety and the Optimal Regimen of VP-102, a Proprietary Drug-Device Product Containing Topical Cantharidin (0.7% w/v) Under Occlusion for the Treatment of Common Warts. Dermatol Ther (Heidelb). 2021 Oct;11(5):1623-1634. doi: 10.1007/s13555-021-00576-y. Epub 2021 Jul 21. PMID 34286459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was originally designed with one- cohort, it was later modified to include two cohorts. Subjects in Cohort 1 completed enrollment prior to beginning enrollment of new Subjects into Cohort 2.
Groups:
- Cohort 1: Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator. utilized a treatment interval of at least 14 days between treatments with longer treatment intervals being allowed depending on a specific patient's clinical response. No paring of lesions was allowed. Subjects were 2 years and older.
- Cohort 2: Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator. Utilized a treatment interval of at least 21 days between treatments with longer treatment intervals being allowed depending on a specific patient's clinical response. Paring of lesions was allowed. Subjects were 12 years and older.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 21 | 35
Completed | 17 | 33
Not Completed | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Study participants enrolled into Cohort 1 were not included in Cohort 2. New subjects were enrolled into Cohort 2.
Groups:
- VP-102 - Cohort 1: Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator.
  Utilized a treatment interval of at least 14 days between treatments with longer treatment intervals being allowed depending on a specific patient's clinical response. No paring of lesions was allowed.
  VP-102 Cantharidin topical film forming solution: VP-102 Cantharidin topical film forming solution. Treatment interval of at least 14 days between treatments.
  VP-102 Applicator: The applicator is used to apply the Study drug.The product is a combination therapy which includes the drug VP-102 and the applicator which is the device.
- VP-102 - Cohort 2: Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator.
  Utilized a treatment interval of at least 21 days between treatments with longer treatment intervals being allowed depending on a specific patient's clinical response. Paring of lesions was allowed.
  VP-102 Cantharidin topical film forming solution: VP-102 Cantharidin topical film forming solution. Treatment interval of at least 21days between treatments.
  VP-102 Applicator: The applicator is used to apply the Study drug.The product is a combination therapy which includes the drug VP-102 and the applicator which is the device.
- Total: Total of all reporting groups
Arm/Group | VP-102 - Cohort 1 | VP-102 - Cohort 2 | Total
Number analyzed (Participants) | 21 | 35 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 8 | 13
  Between 18 and 65 years | 8 | 26 | 34
  >=65 years | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.86 (21.247) | 37.66 (16.435) | 37.75 (18.212)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 22 | 33
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 34 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 16 | 34 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 35 | 56
Baseline wart count [Mean (Standard Deviation); unit: Baseline wart count] | 2.19 (1.569) | 1.65 (1.098) | 1.85 (1.311)

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts (Baseline and New) at the EOS Visit (Day 84)
Description: Cohort 1: Proportion of subjects exhibiting complete clearance of all treatable warts (baseline and new) at the EOS Visit (Day 84).
Time Frame: Treatment Visit Day 1 (Baseline) compared to Day 84 (EOS) Visit.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Participants | 4

2. Primary Outcome: Cohort 2: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts (Baseline and New) at the EOT Visit (Day 84)
Description: Cohort 2: Proportion of subjects exhibiting complete clearance of all treatable warts (baseline and new) at the EOT Visit (Day 84).
Time Frame: Compare Treatment Visit 1 (Baseline) to EOT Visit (Day 84)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Groups:
- VP-102 - Cohort 2: Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator.
  Utilized a treatment interval of 21 days between treatments. Paring of lesions was allowed.
  VP-102 Cantharidin, topical film forming solution: VP-102 Cantharidin topical film forming solution. Treatment interval of at least 21 days between treatments.
  VP-102 Applicator: The applicator is used to apply the Study drug.The product is a combination therapy which includes the drug VP-102 and the applicator which is the device.
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
Participants | 18

3. Secondary Outcome: Cohort 1: Change From Baseline in the Number of Treatable Warts (Baseline and New) at the EOS Visit (Day 84)
Description: Cohort 1: Change from baseline in the number of treatable warts (baseline and new) at the EOS Visit (Day 84).
Time Frame: Change in the number of warts compared at Baseline (Visit 1) to the End of Study Visit (Day 84).
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Number of warts
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Number of warts
  Baseline | 2.19 (1.569)
  End of Treatment Visit | -0.95 (1.658)

4. Secondary Outcome: Cohort 1: Percent Change From Baseline in the Number of Treatable Warts (Baseline and New) at the EOT Visit (Day 84).
Description: Cohort 1: Assessing the percent change from Baseline in the number of treatable warts (Baseline and new) at the EOT visit (Day 84).
Time Frame: Baseline (Visit 1) to End of Treatment Visit (Day 84).
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Percent change | -31.19 (42.776)

5. Secondary Outcome: Cohort 1: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts (Baseline and New) at Visit 2, Visit 3, Visit 4 and Over the Duration of the Study
Description: Cohort 1: Proportion of subjects exhibiting complete clearance of all treatable warts (baseline and new) at Visit 2, Visit 3, Visit 4 and over the duration of the study.
Time Frame: Baseline, Day 14, 28, 42 and 84 (EOS)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Participants
  Complete Clearance Reported at any Visit? | 5
  Complete Clearance Reported at Day 14 | 0
  Complete Clearance Reported at Day 28 | 2
  Complete Clearance Reported at Day 42 | 5
  Complete Clearance Reported at Day 84 (EOS) | 4

6. Secondary Outcome: Cohort 2: Change From Baseline in the Number of Treatable Warts (Baseline and New) at the EOT Visit Day 84)
Description: Cohort 2: Change from baseline in the number of treatable warts (baseline and new) at the EOT Visit Day 84).
Time Frame: Baseline, Day 84 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: change in wart count
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
change in wart count | -0.85 (1.064)

7. Secondary Outcome: Cohort 2: Change From Baseline in the Percent of Treatable Warts (Baseline and New) at the EOT Visit (Day 84)
Description: Cohort 2: Change from baseline in the percent of treatable warts (baseline and new) at the EOT Visit (Day 84).
Time Frame: Baseline (Visit 1) to End of Treatment Visit (Day 84).
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage of change in wart count
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
percentage of change in wart count | -53.79 (55.241)

8. Secondary Outcome: Cohort 2: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts, (Baseline and New), at Visit 2, Visit 3, Visit 4 and Over the Duration of the Study
Description: Cohort 2: Proportion of subjects exhibiting complete clearance of all treatable warts, (baseline and new), at Visit 2, Visit 3, Visit 4 and over the duration of the study.
Time Frame: Baseline, Day 21, 42, 63, and 84 (EOS), 105, 126, and 147
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
Participants
  Complete Clearance Reported at Day 21 (Treatment Visit 2) | 5
  Complete Clearance Reported at Day 42 (Treatment Visit 3) | 7
  Complete Clearance Reported at Day 63 (Treatment Visit 4) | 12
  Complete Clearance Reported at Day 84 (EOT) | 18
  Complete Clearance Reported at Day 105 | 16
  Complete Clearance Reported at Day 126 | 13
  Complete Clearance Reported at Day 147 | 13

9. Other Pre Specified Outcome: Cohort 1:Percent Reduction of All Treatable Warts (Baseline and New) From Baseline at Visit 2, Visit 3, Visit 4 and Over the Duration of the Study.
Description: Cohort 1: Percent change from baseline in the number of treatable warts (Baseline and new) from Baseline at Visit 2, Visit 3, Visit 4 and over the duration of the study.
Time Frame: Baseline, Day 14, 28, 42, and 84 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percent change in number of warts
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Percent change in number of warts
  Treatment Visit 2 Day 14 | -0.79 (3.637)
  Treatment Visit 3 Day 28 | -12.30 (30.462)
  Treatment Visit 4 Day 42 | -29.29 (42.845)
  EOS Day 84 | -31.19 (42.776)

10. Other Pre Specified Outcome: Cohort 1: Change From Baseline in the Number of Treatable Warts (Baseline and New) at Visit 2, Visit 3, Visit 4 and the EOS Visit
Description: Cohort 1: Change from baseline in the number of treatable warts (baseline and new) at Visit 2, Visit 3, Visit 4 and the EOS Visit.
Time Frame: Baseline, Day 14, 28, 42, and 84 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: change in wart count
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
change in wart count
  Treatment Visit 2 | -0.5 (0.218)
  Treatment Visit 3 | -0.43 (1.326)
  Treatment Visit 4 | -0.76 (1.446)
  End of Study | -0.95 (1.658)

11. Other Pre Specified Outcome: Cohort 1: Proportion of Subjects Exhibiting ≥ 50% Clearance of All Treatable Warts (Baseline and New) at the EOS Visit as Compared to Baseline
Description: Cohort 1: Proportion of subjects exhibiting ≥ 50% clearance of all treatable warts (baseline and new) at the EOS visit as compared to baseline.
Time Frame: Compare Treatment Visit 1 (Baseline) to End of Study (Day 84).
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Participants | 7

12. Other Pre Specified Outcome: Cohort 1-Proportion of Subjects Who Respond to Treatment Defined by a ≥ 50% Reduction in Total Wart Area at EOS Compared to Baseline
Description: Cohort 1-Proportion of subjects who respond to treatment defined by a ≥ 50% reduction in total wart area at EOS compared to baseline.
Time Frame: Baseline, Day 14, 28, 42, and 84 (EOS)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Participants | 9

13. Other Pre Specified Outcome: Cohort 1-Proportion of Subjects Exhibiting Reduction of at Least 1 Treatable Wart From Baseline at Visit 2, Visit 3, Visit 4 and at the EOS Visit (Day 84)
Description: Cohort 1-Proportion of subjects exhibiting reduction of at least 1 treatable wart from baseline at Visit 2, Visit 3, Visit 4 and at the EOS Visit (Day 84).
Time Frame: Baseline, Day 14, 28, 42, and 84 (EOS)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 21
Participants
  Reduction of >= 1 Wart from Baseline at any visit? | 9
  Wart Reduction >= 1 Reported at Day 14 (Visit 2) | 1
  Wart Reduction >= 1 Reported at Day 28 (Visit 3) | 4
  Wart Reduction >= 1 Reported at Day 42 (Visit 4) | 8
  Wart Reduction >= 1 Reported at Day 84 (EOS) | 7

14. Other Pre Specified Outcome: Cohort 2: Percent Reduction of All Treatable Warts (Baseline and New) From Baseline at Visit 2, Visit 3, Visit 4 and Over Duration of the Study.
Description: Cohort 2: Intent to Treat population Cohort 2-Percent reduction of all treatable warts (baseline and new) from baseline at Visit 2, Visit 3, Visit 4 and over duration of the study.
Time Frame: Baseline to Treatment Visits 2 (Day 21), 3 (Day 42), 4 (Day 63) through the End of Treatment (Day 84).
Population: ITT population
Measure: Mean (Standard Deviation); unit: percentage of change in wart count
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
percentage of change in wart count
  Day 21 (Treatment Visit 2) | -18.18 (37.119)
  Day 42 (Treatment Visit 3) | -29.85 (41.392)
  Day 63 (Treatment Visit 4) | -37.12 (53.078)
  Day 84 (End of Treatment Visit) | -53.79 (55.241)

15. Other Pre Specified Outcome: Cohort 2: Change From Baseline in the Number of Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4 and the EOT Visit (Day 84)
Description: Cohort 2: Change from baseline in the number of treatable warts (baseline and new) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4 and the EOT Visit (Day 84).
Time Frame: Baseline, Day 14, 28, 42, and 84 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: change in wart count
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
change in wart count
  Day 21 (Treatment Visit 2) | -0.39 (0.998)
  Day 42 (Treatment Visit 3) | -0.48 (0.712)
  Day 63 (Treatment Visit 4) | -0.52 (0.712)
  Day 84 (End of Treatment Visit) | -0.85 (1.064)

16. Other Pre Specified Outcome: Cohort 2: Proportion of Subjects Exhibiting ≥ 50 % Clearance of All Treatable Warts (Baseline and New) at the EOT Visit (Day 84) as Compared to Baseline
Description: Cohort 2: Proportion of subjects exhibiting ≥ 50 % clearance of all treatable warts (baseline and new) at the EOT Visit (Day 84) as compared to baseline.
Time Frame: Baseline to Day 84 (EOT)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
Participants | 19

17. Other Pre Specified Outcome: Cohort 2: Proportion of Subjects Who Respond to Treatment Defined by a ≥ 50% Reduction in Total Wart Area at EOT Compared to Baseline
Description: Cohort 2: Proportion of subjects who respond to treatment defined by a ≥ 50% reduction in total wart area at EOT compared to baseline.
Time Frame: Baseline to EOT (Day 84)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
Participants | 23

18. Other Pre Specified Outcome: Cohort 2: Proportion of Subjects Exhibiting Reduction of at Least 1 Treatable Wart From Baseline at Visit 2, Visit 3, Visit 4 and at the EOT Visit (Day 84)
Description: Cohort 2: Proportion of subjects exhibiting reduction of at least 1 treatable wart from baseline at Visit 2, Visit 3, Visit 4 and at the EOT Visit (Day 84).
Time Frame: Baseline, Day 14, 28, 42, and 84 (EOS)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
Participants
  Day 21 (Treatment Visit 2) | 7
  Day 42 (Treatment Visit 3) | 13
  Day 63 (Treatment Visit 4) | 15
  Day 84 (End of Treatment Visit) | 20

19. Other Pre Specified Outcome: Cohort 2: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts (Baseline and New) at Follow-up Visits on Day 105, Day 126 and Day 147
Description: Cohort 2: Proportion of subjects exhibiting complete clearance of all treatable warts (baseline and new) at follow-up visits on Day 105, Day 126 and Day 147.
Time Frame: Treatment Visit 1 (Baseline) to each follow-up visit Day 105, Day 126 and Day 147.
Measure: Count of Participants; unit: Participants
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
Participants
  Complete Clearance Reported at Day 105 | 16
  Complete Clearance Reported at Day 126 | 13
  Complete Clearance Reported at Day 147 | 13

20. Other Pre Specified Outcome: Cohort 2: Percent Reduction of All Treatable Warts (Baseline and New) From Baseline at Follow-up Visits on Day 105, Day 126 and Day 147
Description: Cohort 2: Percent reduction of all treatable warts (baseline and new) from baseline at follow-up visits on Day 105, Day 126 and Day 147.
Time Frame: Baseline to follow-up visits on Day 105, Day 126 and Day 147
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from Baseline
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
percentage change from Baseline
  Day 105 | -50.91 (54.736)
  Day 126 | -45.61 (52.556)
  Day 147 | -45.61 (52.556)

21. Other Pre Specified Outcome: Cohort 2: Change From Baseline in the Number of Treatable Warts (Baseline and New) at Follow-up Visits on Day 105, Day 126 and Day 147
Description: Cohort 2: Change from baseline in the number of treatable warts (baseline and new) at follow-up visits on Day 105, Day 126 and Day 147.
Time Frame: baseline to Day 105, Day 126 and Day 147
Population: ITT Population
Measure: Mean (Standard Deviation); unit: change in wart count
Arm/Group | VP-102 - Cohort 2
Number analyzed (Participants) | 35
change in wart count
  Day 105 | -0.82 (0.983)
  Day 126 | -0.73 (0.911)
  Day 147 | -0.73 (0.911)

ADVERSE EVENTS:
Time Frame: Cohort 1: Day of first treatment until Day 84 Cohort 2: Day of first treatment until Day 84, 105, 126, 147
Description: Treatment Emergent Adverse Events (TEAEs) are defined as those AEx that occurred after dosing and those existing AEs that worsened during the study. If it cannot be determined whether the AE is treatment emergent due to an incomplete onset date, the AE was considered treatment emergent. Local skin reactions to treatment were recorded as AEs.
Groups:
- Cohort 2: Open label of VP-102 cantharidin topical film forming solution, using the VP-102 applicator. Utilized a treatment interval of 21 days between treatments. Paring of lesions was allowed. Subjects were 12 years and older.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/35
Other Adverse Events (participants affected / at risk) | 20/21 | 32/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=21) | Cohort 2 (N=34)
Application site vesicles (General disorders) | 20 | 27
Application site pain (General disorders) | 20 | 26 — Application site pain
Application site erythema (General disorders) | 13 | 19 — Application site erythema
Application site pruritus (General disorders) | 9 | 16 — Application site pruritus
Application site scab (General disorders) | 8 | 20 — Application site scab
Application site dryness (General disorders) | 6 | 13 — Application site dryness
Application site oedema (General disorders) | 4 | 6 — Application site oedema
Application site discolouration (General disorders) | 1 | 8 — Application site discolouration
Application site exfoliation (General disorders) | 0 | 4 — Application site exfoliation
Application site erosion (General disorders) | 0 | 3 — Application site erosion
Papilloma viral infection (Infections and infestations) | 0 | 3 — Papilloma viral infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is bound to terms and conditions of a Sponsored Clinical Trial Agreement which has strict confidentiality obligations running to Sponsor and broad provisions restricting PI's rights to publish or present any data or Study Results without Sponsor's express review consent and review.

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03487549/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03487549/SAP_001.pdf